CLINICAL TRIAL: NCT02513355
Title: Endostar Treatment of Advanced Non-small Cell Lung Cancer Multi-center Clinical Research
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing NingQi Medicine Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-ENDO-001
Record Dates: First submitted 2015-07-17; First posted 2015-07-31 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer,Endostar
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NP(Changchun marina+cisplatin)+Endostar (Experimental): Patients in this group will be given conventional chemotherapy medicine,NP plan (Changchun marina+cisplatin)recommended by treatment guidelines for Advanced non small cell lung cancer. Endostar 15mg/m2, 21 days per cycle, 4 to 6 cycles;Changchun marina;25mg/m2,d1 and d8,cisplatin 80mg/m2,d1, q21d×4
  Interventions: Biological: Endostar; Drug: Changchun marina; Drug: cisplatin
- TP(Taxol+cisplatin or parapl) +Endostar (Experimental): Patients in this group will be given conventional chemotherapy medicine,TP(Taxol+cisplatin)recommended by treatment guidelines for Advanced non small cell lung cancer.
  Endostar 15mg/m2, 21 days per cycle, 4 to 6 cycles; Taxol;135-175mg/m2,d1,cisplatin or parapl 75mg/m2,d1,q21d×4.
  Interventions: Biological: Endostar; Drug: cisplatin; Drug: Taxol; Drug: parapl

INTERVENTIONS:
Biological: Endostar — Endostar 15mg/m2, 21 days per cycle, 4 to 6 cycles
Drug: Changchun marina — 25mg/m2,d1 and d8,q21d×4
  Arms: NP(Changchun marina+cisplatin)+Endostar
Drug: cisplatin — 80mg/m2,d1, q21d×4
Drug: Taxol — 135-175mg/m2,d1,q21d×4
  Arms: TP(Taxol+cisplatin or parapl) +Endostar
Drug: parapl — AUC=5-6,d1,q21d×4
  Arms: TP(Taxol+cisplatin or parapl) +Endostar

SUMMARY:
Research purpose:

Degree of continuous intravenous pumping Endostar (human recombinant endostatin) combination chemotherapy regimens including cisplatin two medicine first-line treatment of advanced non-small cell lung cancer (with the exception of EGFR/ALK mutations) efficacy and safety.

DETAILED DESCRIPTION:
1.Research purpose: Degree of continuous intravenous pumping Endostar (human recombinant endostatin) combination chemotherapy regimens including cisplatin two medicine first-line treatment of advanced non-small cell lung cancer (with the exception of EGFR/ALK mutations) efficacy and safety.

2.1 main objectives: PFS 2.2 the secondary goal: 2.2. 1 ORR, DCR and OS 2.2. 2 the quality of life 3. The study design 3.1 research nature This is a single arm, multicenter clinical study, is expected to total 100 patients into the group.

Hierarchical factors include: the tumor staging (Ⅲ B vs Ⅳ), ECOG score (0 v 1), gender (male vs female).

3.2 research center and research Proposed by taizhou people's hospital and medical association of jiangsu province tumor chemotherapy and biological branch of the lung cancer group led by several large and medium-sized hospitals in the province of the malignant tumor treatment related department to participate, in accordance with the unified test plan of this research.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation cytology or not in patients undergoing single sputum cytology in the diagnosis of patients with non-small cell lung cancer;
* according to a new IASLC2009 lung cancer TNM stages judged the preious untreated stage IIIB or IV non-small cell lung cancer (with the exception of EGFR/ALK mutations type);
* must have at least one according to the RRECIST version 1.1 standard judgment to evaluate lesions (at least 10 mm, maximum diameter on spiral CT plain CT longest diameter at least 20 mm);
* male or female, age 18 and 75 years old or less or more;
* ECOG PS 0 ~ 1 minute;
* is expected to survive period for 3 months or more,
* enough blood function: absolute neutrophil count (ANC) or 2 x 109 / L and the platelet count 100 x 109 / L or higher acuity 9 g/dL and hemoglobin;
* Liver function enough: upper limit of total bilirubin acuities were normal (ULN); AST and ALT acuities were 2.5 times the upper limit of normal (ULN); Alkaline phosphatase 5 times the upper limit of normal or less (ULN);
* enough renal function, serum creatinine or less normal limit (ULN) or calculated creatinine clearance or 60 mL/min.
* basic normal ecg, had on the body to heal wounds;
* always not received anti-tumor drug therapy, or always only for non metastatic tumor of adjuvant or neoadjuvant chemotherapy, but to study treatment has ended more than six months at the beginning;
* ever had had surgery patients, request to study treatment began to have more than 4 weeks, and the patient has recovered;
* a complete uterus of female in the group within 28 days before the study must have a negative pregnancy test results (except amenorrhea has 24 months). If the pregnancy test from the first time for more than 7 days, is the need for urine pregnancy test validation (within 7 days before the first delivery).
* prior to biological agents, especially e. coli genetically engineered products without severe allergic reactions;
* signed informed consent.

Exclusion criteria

* pregnancy, nursing mothers, or fertility but not women using contraception;
* the existing serious acute infection, and not be controlled; Or fester sex and chronic infection, wound in delay no more;
* the original serious heart disease, including: higher risk of congestive heart failure, unable to control arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension;
* is not easy to control nerve, mental illness or mental disorders, compliance is poor, can't cooperate with accounts and response to treatment; Primary brain tumors or CNS metastases illness did not get a control, has obvious symptoms in cranial hypertension or nerve spirit;
* with bleeding tendency;
* other researchers believe that patients should not participate in this test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
PFS（progression-free survival） | Change from Baseline at the week 6,12, 18 of treatment phase and the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase
  PFS is refers to the patients randomly into group to the date of any objective records of patients with tumor progression or death time.

SECONDARY OUTCOMES:
ORR（Objective Response Rate） | 1 weeks before treatment, Change from Baseline at the week 6,12, 18 of treatment phase and the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase
DCR(disease control rate) | Change from Baseline at the week 6,12, 18 of treatment phase and the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase
OS（overall survival） | Change from Baseline at the week 6,12, 18 of treatment phase and the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase

CONTACTS AND LOCATIONS:
Overall Officials: Han gaohua, PI, Study Chair — China:Taizhou people's hospital
Locations (1):
- Jiangsu Taizhou People's Hospital, Nanjing, Jiangsu, China